CLINICAL TRIAL: NCT03920566
Title: A Pilot Study To Investigate the Effect of ENZAlutamide on the Anti-Xa Levels of Patients Receiving Direct-acting Anticoagulants (DOACS) (ENZA-D)
Brief Title: The Effect of ENZAlutamide on the Anti-Xa Levels of Patients Receiving DOACs
Acronym: ENZA-D
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Pharmacy Research UK (Unknown); University of Brighton (Other)
Responsible Party: Sponsor
Other Study IDs: CCR 5039
Record Dates: First submitted 2019-03-27; First posted 2019-04-19 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Drug Interaction
Keywords: Enzalutamide; Anticoagulant Drugs; P-glycoprotein

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Anti-Xa level — Anti-Xa level taken before commencing enzalutamide and repeated after 4 weeks of treatment

SUMMARY:
This study aims to determine the nature and significance of the theoretical drug interaction between enzalutamide (a drug used to treat prostate cancer) and the direct-acting oral anticoagulant drugs (DOACs). This will be done in two ways: a laboratory study which will take place at the University of Brighton, and a clinical study in which patients will be identified who are currently taking DOACs and are due to start treatment with enzalutamide. The activity of the DOAC will be monitored using anti-Xa levels before and after commencing treatment with enzalutamide.

DETAILED DESCRIPTION:
Enzalutamide is an effective and well-tolerated treatment for advanced prostate cancer. Unfortunately however, enzalutamide can sometimes interact with other medicines that the patient is taking, altering their concentration in the blood-stream. Enzalutamide can do this in two ways: either by increasing the breakdown of a medicine, or by blocking a special protein, called p-glycoprotein, that pumps it out of the body. An example of a medicine whose breakdown is increased by enzalutamide is warfarin. Warfarin is used to prevent, and treat blood clots that have formed in the deep veins of the legs (deep vein thrombosis or DVT) or have become lodged in blood vessels in the lungs (pulmonary embolism or PE). As enzalutamide is known to reduce the effect of warfarin, the manufacturer advises avoiding using the two medicines together. Instead,we can use a new class of medicines called the direct oral anticoagulants, or DOACs.

DOACs have an additional advantage over warfarin in that they do not require regular monitoring with blood tests. We, and other experts in the field believe that there may be a problem using DOACs and enzalutamide together, however scientific evidence suggests that enzalutamide may stop the p-glycoprotein pump from working properly, and alter its ability to pump out a range of medicines. Other evidence suggests that under certain conditions, enzalutamide may actually increase the activity of P-glycoprotein, and reduce the concentration of other medicines in the bloodstream. However, there is no scientific evidence, or evidence from patients, that has looked directly at thecombination of enzalutamide and DOACs together. Because no routine monitoring is carried out with DOACs, we are not sure of the extent of this problem, but the consequences of over or underdosing could be serious.

We have recently generated some preliminary data in our laboratory which has the measured the extent of this interaction, but we need to repeat these experiments before we can draw any firm conclusions from them. In this pilot study, we will explore the potential interaction between enzalutamide and DOACs. First, we will measure the activity of DOACs in patients who are due to start treatment with enzalutamide using a simple, well established blood test. We will then repeat this blood test after the first month of treatment, along with regular blood tests, to determine if there has been a change in the effectiveness of the DOAC. Second, we aim to build uponour laboratory data, and examine whether brief, or prolonged exposure to enzalutamide affects the ability of p-glycoproteinto pump out DOACs.

Our aims are to

1. determine if enzalutamide interacts with DOACs in patients recruited from an advanced prostatecancer clinic
2. understand in greater detail the nature of any interaction between enzalutamide and DOACs in the laboratory
3. assess the feasibility of expanding this study to generate sufficient evidence to make recommendations for clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged > 18 years old
* Diagnosis of castrate resistant metastatic prostate cancer
* Due to commence treatment with enzalutamide
* Currently prescribed edoxaban, rivaroxaban or apixaban
* Calculated CrCl (Cockroft & Gault) > 30ml/min

Exclusion Criteria:

* Patients <18 years old
* Due to stop edoxaban/ rivaroxaban / apixaban during study period (i.e. within 4 weeks of recruitment)
* Currently taking other medicines which induce or inhibit P-gp or increase/reduce the effect of apixaban or rivaroxaban (e.g. verapamil, ketoconazole, itraconazole, voriconazole, ritonavir, clarithromycin, erythromycin (refer to appendix 1 for complete list)
* Currently taking any herbal/complimentary medicines (other than homeopathic products)
* Calculated CrCl (Cockroft & Gault) <30ml/min
* Severe hepatic impairment (Childs-Pugh class C)
* Lacks capacity, including patients with documented dementia (or psychometric marker e.g. Abbreviated Mental Test Score (AMTS) <7/10) or inability to give informed consent for study participation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are currently taking direct-acting oral anticoagulant drugs who are due to start treatment with enzalutamide for the treatment of prostate cancer.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Anti-Xa level | time 0 and time 4 weeks
  Difference between anti-Xa levels taken at two time points (baseline and 4-weeks after commencing enzalutamide)
Efflux ratio (with enzalutamide) | Each experiment will be conducted over a period of <1 day
  Difference in efflux ratio for edoxaban/ rivaroxaban / apixaban in the absence/presence of enzalutamide over a range of concentrations
Efflux ratio (with enzalutamide and positive control) | Each experiment will be conducted over a period of <1 day
  Difference in efflux ratio for edoxaban/ rivaroxaban / apixaban in the presence of enzalutamide and a positive control (e.g. verapamil, whilst ensuring appropriate statistical power)

SECONDARY OUTCOMES:
Bleeding | 4 weeks
  Common Terminology Criteria for Adverse Events (various types of bleeding or hemorrhage are listed. The most appropriate will be selected and graded 1-5 where Grade 1=Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  Grade 2=Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living.
  Grade 3 = Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living.
  Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to adverse event
Bruising | 4 weeks
  A finding of injury of the soft tissues or bone characterized by leakage of blood into surrounding tissues. Graded according to Common Terminology Criteria for Adverse Events grades 1-2 where grade 1=localized or in a dependent area and grade 2 = generalize bruising
Venous Thromboembolism | 4 weeks
  Common Terminology Criteria for Adverse Events (various different thromboembolic events are listed. The most appropriate will be selected and graded 1-5 where Grade 1=Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  Grade 2=Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living.
  Grade 3 = Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living.
  Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Emma Foreman, Principal Investigator — Royal Marsden NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No